CLINICAL TRIAL: NCT00176436
Title: Double-Blind Study of Atomoxetine for Weight Management in Patients Taking Olanzapine or Clozapine
Brief Title: Atomoxetine for Treatment of Weight Gain in Olanzapine or Clozapine Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-21874; F1D-US-X254
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia
Keywords: Weight loss; Support group; Exercise; Atomoxetine
MeSH Terms: conditions — Schizophrenia; Weight Loss; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active (Active Comparator): Atomoxetine titrated up to 120 mg/day by week 8 and continues at 120 mg/day through week 24. Diet support group, group counseling and exercise.
  Interventions: Behavioral: Group counseling and exercise
- Placebo (Placebo Comparator): Placebo medication, diet support group, group counseling and exercise
  Interventions: Behavioral: Diet support group

INTERVENTIONS:
Behavioral: Diet support group — Diet support group weekly and exercise sessions 3 times/week, placebo medication
  Arms: Placebo
Behavioral: Group counseling and exercise — Support group weekly and exercise sessions 3 times/week for 24 weeks
  Arms: active

SUMMARY:
The study investigates the use of Atomoxetine in combination with exercise and a diet support group (Weight Watchers)to treat weight gain associated with Olanzapine or clozapine. All patients must be adults who have been diagnosed with Schizophrenia or Schizoaffective Disorder.

DETAILED DESCRIPTION:
The study is a 6 month double-blind trial of atomoxetine in combination with a Weight Watchers group to help patients lose the weight they have gained taking olanzapine or clozapine. All participants should have been on Olanzapine or clozapine for at least 6 months and gained 7% of baseline weight or have a BMI of 27 or greater. In addition to the group support, participants are provided supervised exercise sessions and medical supervision. Previous studies of the group process alone were successful in helping patients lose weight. It is hoped that the addition of atomoxetine, which is known to cause appetite suppression, will be more effective in helping subjects lose weight. All subjects will receive either atomoxetine or placebo during the 6 month study.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective Disorder
* Taking olanzapine or clozapine for at least 6 months
* Weight gain of 7% over baseline or BMI greater than or equal to 27

Exclusion Criteria:

* Current treatment with methylphenidate, clonidine, tricyclic antidepressants, bupropion and venlafaxine
* Treatment with other medications known to cause weight gain unless weight stable on medication for 6 months
* Current treatment with other medications for weight loss unless weight stable for 6 months
* Mental Retardation
* Alcohol or Substance Dependence within the last 6 months
* Pregnancy
* Alcohol or Substance Abuse within the lat month
* Uncontrolled hypertension defined as a blood pressure exceeding 140/90 on three consecutive readings despite adequate treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Patricia Ball, R.N.,C.,M.S., Principal Investigator — University of Maryland Baltimore Maryland Psychiatric Research Center
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- [Result] Ball MP, Warren KR, Feldman S, McMahon RP, Kelly DL, Buchanan RW. Placebo-controlled trial of atomoxetine for weight reduction in people with schizophrenia treated with clozapine or olanzapine. Clin Schizophr Relat Psychoses. 2011 Apr;5(1):17-25. PMID 21459735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from 2004 until March, 2008. Participants were recruited from the Maryland Psychiatric Research Center Outpatient Research Program and local community mental health centers.
Pre-assignment Details: There was a 2-week evaluation period during which time a diet and exercise program was implemented. All participants then began the double-blind treatment phase of the study. No participants were excluded unless the were taking an excluded medication. 40 participants were enrolled into active participation; 37 participants started treatment.
Groups:
- Active: Atomoxetine titrated up to 120 mg/day by week 8 and continues at 120 mg/day through week 24.
- Placebo: Placebo medication, diet support group weekly and exercise sessions 3 times/week
Period: Overall Study
Arm/Group | Active | Placebo
Started | 20 | 17
Completed | 14 | 12
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (8.4) | 46.1 (9.4) | 46.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight
Description: Weight loss was measured each week over the 24 week study period. Intent to treat analyses of treatment effects on the primary outcome (weight) were conducted using all observed weight measurements from all participants with post-baseline weight measurements, using the mixed model for unbalanced repeated measures ANOVA. This model summarizes change in weight for each participant by the average change in weight per week (slope) over 24 weeks, and compares these slopes between the two groups.
Time Frame: Weekly for 24 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Active | Placebo
Number analyzed (Participants) | 20 | 17
kilograms | 1.7 (1.4) | 2.1 (1.4)

2. Secondary Outcome: Secondary Outcomes Are Improvement in Cognitive Impairments, Since Atomoxetine is Used for Treatment of ADHD and is Known to Improve Cognitive Function.
Time Frame: 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Vital Signs
Time Frame: Weekly for 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Chemistry Panel
Time Frame: baseline, 10 weeks and 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Weekly questionnaire assessing potential side effects
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 2 | 1
Other Adverse Events (participants affected / at risk) | 5 | 4
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Active | Placebo
Hypotension (Cardiac disorders) | 1/20 | 0/17
Extreme Sedation (General disorders) | 1/20 | 0/17
Chest Pain (Cardiac disorders) | 0/20 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Active | Placebo
Dizziness (Vascular disorders) | 1/20 | 0/17
Slurred speech (Nervous system disorders) | 1/20 | 0/17
Abnormal ECG (Cardiac disorders) | 1/20 | 0/17
Hypotension (Cardiac disorders) | 1/20 | 0/17
Nervousness (Psychiatric disorders) | 1/20 | 0/17
Hypertension (Cardiac disorders) | 0/20 | 1/17
Cough (Respiratory, thoracic and mediastinal disorders) | 0/20 | 1/17
Abnormal SGOT and SGPT (Blood and lymphatic system disorders) | 0/20 | 1/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes